CLINICAL TRIAL: NCT04406532
Title: Home Based Covid-19 Rehabilitation Program: Pilot Clinical Trial
Brief Title: Home-Based Covid-19 Rehabilitation Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never started due to recruitment difficulties. The rates of COVID infections in the recruitment area declined significantly.
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Joe Verghese, Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-11535
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Covid-19
Keywords: rehabilitative medicine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PT-Pal (Experimental): Participants randomized to the 14-day intervention arm will receive exercise instructions via PT-Pal. The Pt-Pal is a mobile health technology used to facilitate communication between the Care Team and patients, by allowing the team to send from their web-portal, exercise routines, surveys and educational material to the patient's mobile device. The PT-Pal app then captures the patient activity adherence, and reports those results back to the team including a graphical summary about patients' condition and activity. Clinicians can send/receive HIPAA-secure messages with patients. The app was designed to work with intermittent data connectivity typically found in mobile networks by switching between store-and-forward and real-time mode of connectivity to ensure data delivery.
  Interventions: Behavioral: PT-Pal
- Self-guided exercises (Active Comparator): Participants randomized to the 14-day control arm will be instructed by research staff on how to use the exercise manual provided at the time of their screening.
  Interventions: Behavioral: Self-guided exercises

INTERVENTIONS:
Behavioral: PT-Pal — Participants will be guided through an exercise program in the PT-Pal app. The program is stratified into 3 levels. Participants begin with Level 1 exercises to prevent atelectasis, strengthen inspiratory and expiratory muscles. Gradually exercises to stretch limb and chest wall muscles, build sitting tolerance and to improve transfer ability are added. These exercises can improve respiratory vital capacity. Level 2 focuses on sitting tolerance, strengthening limb and accessory muscles of breathing. Level 3 focuses on standing balance, large muscle strengthening, and building cardiopulmonary endurance.
  Each exercise is done 2-3 times, and gradually increased to a complete set of 8. Each set is then repeated 2-3 per day, building up tolerance and fitness. Duration of session varies from 10 min initially up to 45 min later depending on fitness.
  Arms: PT-Pal
Behavioral: Self-guided exercises — Participants will use the exercise manual to guide the exercise program. The program is stratified into 3 levels. Participants begin with Level 1 exercises to prevent atelectasis, strengthen inspiratory and expiratory muscles. Gradually exercises to stretch limb and chest wall muscles, build sitting tolerance and to improve transfer ability are added. These exercises can improve respiratory vital capacity. Level 2 focuses on sitting tolerance, strengthening limb and accessory muscles of breathing. Level 3 focuses on standing balance, large muscle strengthening, and building cardiopulmonary endurance.
  Each exercise is done 2-3 times, and gradually increased to a complete set of 8. Each set is then repeated 2-3 per day, building up tolerance and fitness. Duration of session varies from 10 min initially up to 45 min later depending on fitness.
  Arms: Self-guided exercises

SUMMARY:
Our aim is to conduct a pilot single-blind randomized controlled trial to examine the preliminary efficacy of a 14 day app-based pulmonary and mobility focused rehabilitation program (intervention arm) versus a self-guided exercise program (active control arm) on pulmonary and functional outcomes in 100 patients tested for COVID-19 infection and isolated at home.

DETAILED DESCRIPTION:
As of April 20, 2020, there had been over 2.4 million confirmed cases of coronavirus disease 2019 (COVID-19) reported globally; 759,786 cases in USA. Triage protocols have been developed to prioritize individuals for COVID-19 testing based on exposure or symptoms. Due to the high demand for screening, the turnaround time for results in our area varies from 5-6 days. While current estimates suggest that 80% of individuals will have mild illness, there is no reliable way to predict course. Also some patients may rapidly deteriorate a week after illness onset. No proven preventive or therapeutic options are yet available for individuals with mild symptoms who are tested for COVID-19 infection, and asked to self-isolate themselves at home while awaiting results.

COVID-19 is mainly a respiratory disease. Complications such as pneumonia and acute respiratory distress syndrome (ARDS) are among its most dreaded complications, and major contributors to Intensive Care Unit admissions and mortality. Early studies show that dyspnea occurs at a median of 6 days after initial symptom onset, which can progress to ARDS at a median of 12 days after onset. Hence, there is a window of 3-4 days after symptom onset (corresponds to the time individuals typically wait for test results) that interventions could be applied to prevent progression. Pulmonary and functional rehabilitation has proven validity in preventing worsening of pulmonary and physical function in respiratory diseases. But the utility of rehabilitation has not yet been established in the COVID-19 patient population.

Based on our research in frail older adults and input from experts, the investigators recently developed and published an innovative stratified self-guided care and exercise manual for patients with COVID-19 infection to improve pulmonary function and prevent immobility. The investigators build on this experience to test the efficacy of a telephone-based app (PT-Pal™) version of this pulmonary and mobility focused rehabilitation program. The PT-Pal is a validated cloud-based patient engagement platform that enables management of patient care by sending treatment plans, surveys and reminders to the patient's mobile device using HIPAA compliant secure messaging.

Our aim is to conduct a pilot single-blind randomized controlled trial in 100 patients tested for COVID-19 infection and isolated at home who will be randomized into either a 14 day PT-Pal pulmonary and mobility focused rehabilitation program or a self-guided exercise group. Compared to participants in the active control group, the investigators hypothesize that participants in the PT-Pal program will show lesser declines in self-reported pulmonary (St George's Respiratory questionnaire) and physical function (AM-PAC basic mobility questionnaire) due to greater participation and adherence rates. The investigators will test at baseline, day and day 14 to determine trajectories in both groups. All outcomes will be collected remotely as social distancing precludes in-person testing. At our recruitment site, 40-45% of individuals tested for COVID-19 had a positive result, but given current delays in obtaining results (5-6 days), the investigators will enroll participants before knowing their COVID-19 status.

The investigators will also examine the following secondary outcomes obtained remotely: Pulmonary function (breath holding and peak flow), Physical function (5 times sit to stand test), Health events (Emergency Room visits, hospitalizations), Psychological (anxiety/depressive symptoms), and Feasibility metrics (sessions completed).

Our pilot clinical trial will build the evidence base for a rehabilitative approach to be applied alongside emerging therapies to ameliorate the devastating pulmonary and physical function declines seen in COVID-19 infection. It can be implemented in the time window between presentation and development of severe symptoms in the large population of adults awaiting test results in the community. Our approach can also apply to COVID-19 patients such as those discharged from hospitals or healthcare workers furloughed home due to disease exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older.
2. Symptoms suggestive of Covid-19 infection (fever, cough, chest discomfort or loss of smell/taste).
3. Covid-19 screening done.
4. Ambulatory without assistive devices (such as cane or walker).
5. Access to PT-Pal app via cellular phone, iPad or computer (e.g. Zoom™).

Exclusion Criteria:

1. Severe symptoms requiring referral to the Emergency Department.
2. Contraindications to exercise (cardiac disease such as diagnosed arrhythmias, on home oxygen, or end stage organ failure).
3. Known history of poorly controlled diabetes or hypertension.
4. Active neurological or psychiatric illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary function (St George's Respiratory questionnaire: SGRQ) | baseline, at day 7 and at day 14
  The SGRQ is a valid instrument for measuring pulmonary function in patients with respiratory disease, with a total score and scores for symptom, physical activity, and impact domains (range 0 to 100; higher scores worse). The minimum clinically important difference is 4 points. The questionnaire has excellent reliability and validity compared to gold standard pulmonary function tests.
Change in physical function (Activity Measure for Post-Acute Care: AM-PAC) | baseline, at day 7 and at day 14
  The AM-PAC was developed to examine basic mobility and daily activity functional activities important to adults. It is a validated measure of patient-reported functional limitation in 3 domains: basic mobility, daily activities, and applied cognition. It is endorsed by the National Quality Forum as a functional status quality metric.

SECONDARY OUTCOMES:
Change in pulmonary function (Sabrasez single breath count) | baseline, at day 7 and at day 14
  Patient asked to take a deep breath while at rest and to hold it (Normal >25 s). Test monitored by video (Zoom, PT-Pal).
Change in pulmonary function (Peak flow tests) | baseline, at day 7 and at day 14
  Participants will be given a peak flow meter at recruitment, and taught how to use it by research staff over video.
Change in physical function (5 times site to stand test) | baseline, at day 7 and at day 14
  This timed test assesses strength, balance and endurance. Test monitored by video (Zoom, PT-Pal).
Health events (emergency room visits and hospitalizations) | baseline to day 14
  Self-report or information from medical staff.
Change in psychological measures (Beck Anxiety Inventory: BAI) | baseline, at day 7 and at day 14
  Anxiety symptoms reported on the BAI. Higher scores indicate more anxiety.
Change in psychological measures (Center for Epidemiologic Studies Depression Scale: CES-D) | baseline, at day 7 and at day 14
  Depressive symptoms reported on the CES-D. Higher score indicate more depressive symptoms.
Feasibility (Adherence) | baseline to day 14
  Number of sessions completed using app in the intervention arm. Controls periodically interviewed.
Feasibility (Acceptability) | baseline to day 14
  Survey of satisfaction with exercise programs.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Verghese, MBBS, Principal Investigator — Albert Einstein College of Medicine; Anne F Ambrose, MD, Principal Investigator — Albert Einstein College of Medicine

IPD SHARING:
Plan to Share IPD: No